CLINICAL TRIAL: NCT04852341
Title: Study on the Difference of Preoperative Related Parameters in Children With or Without Microcornea Within Less Than One Year Old
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Deputy Dean, Wenzhou Medical University
Other Study IDs: Microcornea
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Microcornea Within One Year of Age
MeSH Terms: interventions — Tonometry, Ocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Corneal horizontal diameter ≤9.00mm group
  Interventions: Device: Collect ocular biological parameters including age, corneal diameter, eye axis, intraocular pressure, steep&flat axis of corneal curvature, corneal thickness, lens thickness, anterior chamber depth
- Corneal horizontal diameter 9.00mm~9.50mm group
  Interventions: Device: Collect ocular biological parameters including age, corneal diameter, eye axis, intraocular pressure, steep&flat axis of corneal curvature, corneal thickness, lens thickness, anterior chamber depth
- Corneal horizontal diameter 9.50mm~10.00mm group
  Interventions: Device: Collect ocular biological parameters including age, corneal diameter, eye axis, intraocular pressure, steep&flat axis of corneal curvature, corneal thickness, lens thickness, anterior chamber depth
- Corneal horizontal diameter >10.00mm group
  Interventions: Device: Collect ocular biological parameters including age, corneal diameter, eye axis, intraocular pressure, steep&flat axis of corneal curvature, corneal thickness, lens thickness, anterior chamber depth

INTERVENTIONS:
Device: Collect ocular biological parameters including age, corneal diameter, eye axis, intraocular pressure, steep&flat axis of corneal curvature, corneal thickness, lens thickness, anterior chamber depth — observation

SUMMARY:
This subject is mainly to study difference of Congenital cataract preoperative related parameters in children with or without Microcornea within Less than one year old. A total of 186 eyes of 117 people were collected with relevant ocular biological parameters, including age, horizontal diameter of the cornea, Eye axis, intraocular pressure, steep axis of corneal curvature, flat axis of corneal curvature, corneal thickness, lens thickness, anterior chamber depth. At present, because the definition of patients with small cornea is not clear enough, the study subjects are divided into 4 groups according to the horizontal corneal diameter of 9.0mm, 9.5mm, and 10.0mm, namely ≤9.0mm group, 9~9.5mm group, 9.5~10.0mm group and The >10.0mm group compares the differences between each other, and tries to provide a reference for the diagnosis of children with small cornea at a young age.

ELIGIBILITY:
Inclusion Criteria:

* Congenital cataract children with or without Microcornea within Less than one year old
* Complete collection of eye biological parameters before the first-stage Congenital cataract surgery
* The nutritional status and development of the included subjects have no obvious defects

Exclusion Criteria:

* congenital persistent pupilary membrane
* lens sublaxation or lens dislocotion
* Marfan syndrome
* Down's Syndrome
* Peters abnormality
* Fevr
* history of obvious eye trauma
* obvious macula
* long-term (local or systemic) use of glucocorticoids.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: From May 2015 to December 2020,Congenital cataract children with or without Microcornea within one year of age attending the Eye Optometry Hospital of Wenzhou Medical University
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
horizontal diameter of the cornea | 2015.5.1-2020.12.1
  Use a ruler to measure during surgery

SECONDARY OUTCOMES:
age | 2015.5.1-2020.12.1
Eye axis | 2015.5.1-2020.12.1
  A-type ultrasonic measuring instrument
intraocular pressure | 2015.5.1-2020.12.1
  i care handheld tonometer
steep axis of corneal curvature | 2015.5.1-2020.12.1
  Handheld eye curvature measuring instrument
flat axis of corneal curvature | 2015.5.1-2020.12.1
  Handheld eye curvature measuring instrument
corneal thickness | 2015.5.1-2020.12.1
  Handheld corneal thickness measuring instrument
lens thickness | 2015.5.1-2020.12.1
  A-type ultrasonic measuring instrument
anterior chamber depth | 2015.5.1-2020.12.1
  SS-OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Wenzhou Medical University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Zhang H, Chen Z, He K, Chang P, Zhao Y, Huang X, Li J, Jin Z, Zhao YE. Unique presentation of congenital cataract concurrent with microcornea, microphthalmia plus posterior capsule defect in monozygotic twins caused by a novel GJA8 mutation. Eye (Lond). 2019 Apr;33(4):686-689. doi: 10.1038/s41433-018-0277-y. Epub 2018 Nov 29. No abstract available. PMID 30498267
- [Background] Matalia J, Shirke S, Shetty KB, Matalia H. Surgical Outcome of Congenital Cataract in Eyes With Microcornea. J Pediatr Ophthalmol Strabismus. 2018 Jan 1;55(1):30-36. doi: 10.3928/01913913-20170703-13. Epub 2017 Oct 9. PMID 28991349
- [Background] Liu T, Zhang M, Xu B, Wang W, Lee J, Gao Y, Zhang X. Evaluation of the safety of sclerotomy incision in patients with choroidal colobomas with/without associated microcornea. Retina. 2014 Nov;34(11):2300-5. doi: 10.1097/IAE.0000000000000227. PMID 25011027
- See also: Evaluation of the safety of sclerotomy incision in patients with choroidal colobomas with/without associated microcornea — https://pubmed.ncbi.nlm.nih.gov/25011027/
- See also: Surgical Outcome of Congenital Cataract in Eyes With Microcornea. J Pediatr Ophthalmol Strabismus. — https://pubmed.ncbi.nlm.nih.gov/28991349/
- See also: Unique presentation of congenital cataract concurrent with microcornea, microphthalmia plus posterior capsule defect in monozygotic twins caused by a novel GJA8 mutation. — https://pubmed.ncbi.nlm.nih.gov/30498267/